CLINICAL TRIAL: NCT01195376
Title: A Phase I Study of BEZ235, Administered Orally in Adult Japanese Patients With Advanced Solid Tumors
Brief Title: A Study of BEZ235 in Adult Japanese Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBEZ235A1101
Record Dates: First submitted 2010-09-02; First posted 2010-09-06 (Estimated); Last update posted 2020-12-09 (Actual); Status verified 2016-04

CONDITIONS: Advanced Solid Tumor
Keywords: PI3K; mTOR; Advanced solid tumor
MeSH Terms: interventions — dactolisib

ARMS (2):
- BEZ235 Dose Escalation once daily (Experimental): oral BEZ235 once daily (q.d.)
  Interventions: Drug: BEZ235
- BEZ Dose escalation twice daily (Experimental): oral BEZ235 twice daily (b.i.d.)
  Interventions: Drug: BEZ235

INTERVENTIONS:
Drug: BEZ235

SUMMARY:
In this study, BEZ235 will be administered to adult patients with advanced solid tumors whose disease has progressed despite standard therapy or for whom no standard therapy exists. The trial will confirmed the safety and tolerability and determine the MTD of BEZ235 in Japanese patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically-confirmed, advanced unresectable solid tumors who have progressed on (or not been able to tolerate) standard therapy or for whom no standard anticancer therapy exists.
2. At least one measurable lesion as defined by RECIST criteria for solid tumors.
3. Age ≥ 20
4. Eastern Cooperative Oncology Group Performance Status (ECOG P.S.) of ≤ 2
5. Life expectancy of ≥ 12 weeks
6. Patients must have the laboratory values Patients in the expansion part of this study have to meet the following criteria in addition to the criteria described above.
7. Availability of a representative tumor tissue specimen (either archival tumor or fresh tumor biopsy) for pre-screening.
8. Patients whose molecular status proved to meet the criteria (PIK3CA mutation/amplification and/or PTEN mutation and/or low/null PTEN expression) during pre-screening.

Exclusion Criteria:

1. Patients who have brain metastases or who have signs/symptoms attributable and have not been assessed with radiologic imaging to rule out the presence of brain metastases
2. Patients with any peripheral neuropathy ≥ CTCAE grade 2
3. Patients with unresolved diarrhea ≥ CTCAE grade 2
4. Patients with a history of photosensitivity reactions to other drugs
5. Women of child-bearing potential who are pregnant or breast feeding or adults of reproductive potential not employing an effective method of birth control. Barrier contraceptives must be used throughout the trial in both sexes. Women of child-bearing potential, defined as sexually mature women who have not undergone a hysterectomy or who have not been naturally postmenopausal for at least consecutive 1 years (i.e., who has had menses any time in the preceding consecutive 2 years), must have a negative serum pregnancy test ≤ 7 days prior to starting BEZ235.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2010-10; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
To establish Maximum tolerate dose (MTD) | Every week

SECONDARY OUTCOMES:
Safety assessed by type, frequency and severity of adverse events | Every week
Efficacy assessed by RECIST | Every 2 months
To characterize the PK profiles | Every 2 weeks
To assess the biomarkers | Every 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Japan (2):
  - Novartis Investigative Site, Kobe, Hyōgo
  - Novartis Investigative Site, Yufu, Oita Prefecture

REFERENCES:
- [Derived] Toyoda M, Watanabe K, Amagasaki T, Natsume K, Takeuchi H, Quadt C, Shirao K, Minami H. A phase I study of single-agent BEZ235 special delivery system sachet in Japanese patients with advanced solid tumors. Cancer Chemother Pharmacol. 2019 Feb;83(2):289-299. doi: 10.1007/s00280-018-3725-2. Epub 2018 Nov 16. PMID 30446785
- See also: Results for CBEZ235A1101 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=11645